CLINICAL TRIAL: NCT06769659
Title: A Single-center, Double-blind, Placebo-controlled Crossover Study Evaluating NPT 2042 Versus Placebo in Subjects Aged 16-75 Years With Genetic Generalized Epilepsy (GGE) and Absence Seizures
Brief Title: A Study Evaluating NPT 2042 Versus Placebo in Subjects Aged 16-75 Years With Genetic Generalized Epilepsy (GGE) and Absence Seizures
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroPro Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NPT 2042 CL-200
Record Dates: First submitted 2024-12-23; First posted 2025-01-10 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Epilepsy, Generalized; Epilepsy, Absence
MeSH Terms: conditions — Epilepsy, Generalized; Epilepsy, Absence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NPT 2042 80mg (Active Comparator): NPT 2042 80mg BID
  Interventions: Drug: NPT 2042; Other: Placebo
- Placebo (Placebo Comparator): Matching placebo for active comparator
  Interventions: Drug: NPT 2042; Other: Placebo

INTERVENTIONS:
Drug: NPT 2042 — NPT 2042 is a new drug being developed as an anti-seizure treatment
Other: Placebo — Placebo Comparator

SUMMARY:
This study will compare the effect of NPT 2042 and placebo in subjects with GGE on the frequency and duration of electroencephalographic absence seizures, separated by a 14-day washout period. The study will be a single-center, double-blind, crossover study with subjects receiving either NPT 2042 80 mg BID orally or matching placebo BID in each of two treatment periods.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is capable of and provides consent/assent, and the study participant's parent/legal representative/caregiver provides signed informed consent for minor study participants, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF)
2. Subject is aged 16-75 years at the time of consent/assent
3. Subject is diagnosed with genetic generalized epilepsy with absence seizures (consistent with the International League Against Epilepsy (ILAE) Classification of Seizures (2017))
4. Subject has electroencephalogram (EEG) evidence of bilateral synchronous generalized paroxysmal spike-wave (2.5 Hz to 6 Hz) bursts lasting 3 seconds or more at least 4 times on the screening 72-hour ambulatory EEG.
5. Subject has been on a stable dose of at least one antiseizure medication (ASM) for at least 30 days. Vagal nerve stimulation at stable settings (for at least 30 days before screening), without use of the magnet, is also acceptable.
6. Subject has normal cognition and no clinically significant abnormalities on neurological examination at screening in the opinion of the Investigator
7. Subject is in otherwise good health (with the exception of epilepsy), as determined by the investigator, and as documented in the medical history, physical examination, and screening laboratory investigations
8. Subject has a body mass index (BMI) between 18 and 40 kg/m2 inclusive, at screening
9. Female subjects of child-bearing potential and all men agree to use of highly effective methods of contraception during the study and for 28 days after last dose of study drug
10. Subject (and parent/caregiver, if applicable) is able to communicate with the investigator and to understand and comply with all study requirements, including the clinic visit schedule

Exclusion Criteria:

1. Subject has metabolic or mitochondrial encephalopathies, seizures associated with structural abnormalities, or infection-related seizures.
2. Subject has a developmental epileptic encephalopathy (e.g. Lennox-Gastaut syndrome)
3. Subject has a history of convulsive status epilepticus within the past year.
4. Subject has a history of surgical intervention for treatment of epilepsy
5. Subject has a history of nonepileptic seizures (e.g., metabolic, structural, or paroxysmal non epileptic seizures)
6. Subject has severe intellectual disability, severe autism spectrum disorder, or severe developmental disorder such that the subject cannot consent or assent to participate or cannot cooperate with the study procedures
7. Female subject who is pregnant or lactating
8. Subject has any clinically significant laboratory abnormality which, in the opinion of the investigator, will exclude the subject from the study
9. Subject has an active CNS infection, demyelinating disease, degenerative neurological disease, or any CNS disease deemed to be progressive during the course of the study that may confound the interpretation of the study results
10. Subject has any clinically significant psychiatric illness, psychological or behavioral problems which, in the opinion of the investigator, would interfere with the subject's ability to participate in the study, including but not limited to the following:

    1. Subject has active suicidal ideation prior to study entry as indicated by a positive response ("yes") to either Question 4 or Question 5 of the Columbia Suicide Severity Rating Scale (C-SSRS)
    2. Study participant has a lifetime history of suicide attempt (including an active attempt, interrupted attempt, or aborted attempt)
11. Subject is suffering from clinically significant active liver disease, porphyria or has a family history of severe hepatic dysfunction indicated by abnormal liver function tests greater than three times the upper limit of normal (AST and ALT)
12. Subject has a DSM-V diagnosis of alcohol or drug abuse, or drug addiction within the past 12 months
13. Subject has participated in any other trials involving an investigational product or device within 30 days of screening or longer, as required by local regulations
14. Subject is currently using prohibited medications or products
15. Subject is unable to complete ingestion of four placebo SGCs with a minimum of eight ounces of water at screening
16. Subject (and parent/caregiver, if applicable) has daily commitments during the study duration that would interfere with attending all study visits
17. Positive urine drug test for substance of abuse or illegal recreational substances at screening

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Mean and median across subjects of the within subject difference in percent change from treatment period baseline of the frequency of absence seizures | Up to 12 weeks
  Mean and median across subjects of the within subject difference in percent change from treatment period baseline of the frequency of absence seizures (defined as 2.5-6 Hz spike-wave bursts lasting greater than 3 seconds) between NPT 2042 and placebo.

SECONDARY OUTCOMES:
Mean and median across subjects of the within subject difference between NPT 2042 and placebo on absence seizures | Up to 12 weeks
  Mean and median across subjects of the within subject difference between NPT 2042 and placebo on absence seizures (defined as 2.5-6 Hz spike-wave bursts lasting greater than 3 seconds) average duration.
Mean and median across subjects of the within subject categorical difference in percent change between NPT 2042 and placebo of the frequency of absence seizure | Up to 12 weeks
  Mean and median across subjects of the within subject categorical difference in percent change between NPT 2042 and placebo of the frequency of absence seizure (defined as 2.5-6 Hz spike wave bursts lasting greater than 3 seconds) using the following categories:
  * <10 seconds
  * 10-20 seconds
  * >20 seconds
The proportion of NPT 2042- vs. placebo-treated subjects meeting the study specific response criteria | Up to 12 weeks
  The proportion of NPT 2042- vs. placebo-treated subjects meeting the following response criteria:
  * ≥50% decrease in endpoint seizure frequency compared to treatment period baseline
  * ≥75% decrease in endpoint seizure frequency compared to treatment period baseline
  * Seizure freedom
The mean change from Baseline across subjects of the within subject difference between NPT 2042 and placebo on the Quality of Life in Epilepsy Questionnaire (QOLIE-31-P) | Up to 12 weeks
  The mean change from Baseline across subjects of the within subject difference between NPT 2042 and placebo on the Quality of Life in Epilepsy Questionnaire (QOLIE-31-P)
The mean change from Baseline in the Digit Symbol Substitution Test | Up to 12 weeks
  The mean change from Baseline in the Digit Symbol Substitution Test following treatment with NPT 2042 compared to placebo
The mean change from Baseline in the Epworth Sleepiness Scale | Up to 12 weeks
  The mean change from Baseline in the Epworth Sleepiness Scale following treatment with NPT 2042 compared to placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trials, Inc. (CTI), Little Rock, Arkansas, United States